CLINICAL TRIAL: NCT07085143
Title: An Exploratory Randomized, Double-blind, Placebo-controlled Study on Compound Ciwujia Granules in the Treatment of Depression (Heart-Spleen Deficiency Syndrome)
Brief Title: Clinical Study of Compound Ciwujia Granules in the Treatment of Depression
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Heilongjiang Quanle Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-34
Record Dates: First submitted 2025-06-20; First posted 2025-07-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Depression - Major Depressive Disorder; Depression Disorders
Keywords: Compound Ciwujia Granules; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): 1. Take placebo twice daily for 8 weeks;
  2. Continue concomitant SSRI medication therapy throughout the treatment period
  Interventions: Drug: placebo
- intervention group (Experimental): 1. Take Compound Ciwujia Granules twice daily for 8 weeks;
  2. Continue concomitant SSRI medication therapy throughout the treatment period;
  Interventions: Drug: Compound Ciwujia Granules

INTERVENTIONS:
Drug: Compound Ciwujia Granules — Take Compound Ciwujia Granules or placebo twice daily for 8 weeks; Continue concomitant SSRI medication therapy throughout the treatment period;
  Arms: intervention group
Drug: placebo — 1. Take placebo twice daily for 8 weeks;
  2. Continue concomitant SSRI medication therapy throughout the treatment period;
  Arms: control group

SUMMARY:
The purpose of this clinical trial is to evaluate the therapeutic efficacy and safety of Compound Ciwujia Granules in treating depression disorder (heart-spleen deficiency syndrome). The study primarily aims to address the following key questions:

* Can Compound Ciwujia Granules effectively alleviate depressive symptoms in patients with heart-spleen deficiency syndrome?
* What adverse reactions might participants experience while taking Compound Ciwujia Granules? Researchers will compare Compound Ciwujia Granules to a placebo (a look-alike substance that contains no drug) to see if Compound Ciwujia Granules works to treat depression disorder.

Participants are required to complete the following procedures:

1. Take Compound Ciwujia Granules or placebo twice daily for 8 weeks;
2. Continue concomitant SSRIs throughout the treatment period;
3. Return to the hospital for scheduled assessments at Week 4 and Week 8;
4. Complete a 4-week follow-up period after the 8-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) diagnostic criteria for major depressive disorder (MDD) and the depressive episode criteria of the Mini-International Neuropsychiatric Interview (M.I.N.I.);
* Fulfills Traditional Chinese Medicine (TCM) diagnostic criteria for heart-spleen deficiency syndrome
* HAMD-17 (17-item Hamilton Depression Rating Scale) total score: 8-24;
* HAMA (Hamilton Anxiety Rating Scale) score ≤21;
* Outpatient participants aged 18-65 (inclusive) of either sex;
* Education level ≥ junior high school, capable of completing self-assessment scales;
* Currently on a stable dose of one SSRI for ≥6 weeks, with a CGI-GI (Clinical Global Impression - Global Improvement) score ≥4 at screening and baseline;
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Prior diagnosis or medical history of: organic mental disorder-related depression, clinically significant neurological diseases (e.g., epilepsy, encephalopathy), any neurodegenerative disorders, moderate/severe head trauma or other neurological conditions affecting CNS function;
* Current DSM-5-diagnosed psychiatric disorders (other than MDD), including:

Schizophrenia spectrum/other psychotic disorders, Bipolar and related disorders, Anxiety disorders, OCD, or somatic symptom disorders, Substance-related/addictive disorders (excluding caffeine/nicotine), Positive urine drug screen at screening;

* Suicide risk, defined as: history of suicide attempt, investigator-assessed current significant risk, any "Yes" response to C-SSRS Items 1-5;
* Severe systemic diseases, including: significant cardiac, hepatic, or renal dysfunction, ALT/AST >1.5× upper limit of normal (ULN);
* Pregnancy/lactation, or women of childbearing potential not using effective contraception;
* Acute/chronic conditions within 1 month: Infectious/autoimmune diseases, allergies, cancer, or stroke;
* Participation in other drug trials within 1 month;
* History of:psychosurgery, deep brain stimulation (DBS), electroconvulsive therapy (ECT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The change rate of Hamilton Depression Rating Scale-17#HAMD-17# after treatmen | From enrollment to the end of the treatment at 8 weeks
  Reduction rate = (Baseline HAMD-17 score - Week 4 HAMD-17 score) / Baseline HAMD-17 score. A HAMD-17 response rate ≥50% is defined as an effective treatment

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale#HAMA | From enrollment to the end of treatment at 8 weeks
  HAMA scale is used to assess the severity of anxiety symptoms in patients with neurotic disorders and other conditions. Previous studies have reported good reliability and validity for this scale. The scores from all 14 items are summed to give a total score, which indicates the overall severity of anxiety: < 17: Mild severity; 18-24: Mild to moderate severity; 25-30: Moderate to severe severity.
Pittsburgh sleep quality index#PSQI# | From enrollment to the end of the treatment at 8 weeks
  PSQI is used to assess sleep quality over the past month. It is suitable for evaluating sleep quality in patients with sleep disorders and mental disorders, as well as in the general population. The total score ranges from 0 to 21 points. A total score of >7 is commonly used as the cutoff threshold for determining the presence of subjective sleep problems.
Treatment Emergent Symptom Scale#TESS# | From enrollment to the end of treatment at 8 weeks
  Among comparable scales, it provides the most comprehensive item coverage-assessing both common adverse symptoms/signs and multiple laboratory findings. The Treatment Emergent Symptom Scale (TESS) requires clinicians to evaluate each symptom across three dimensions: Severity, Relationship to Intervention, and Action Taken.
  Severity is rated on a 0-4 scale:
  0. = Absence of the symptom;
  1. = Occasional presence of the symptom;
  2. = Mild severity, no impairment to routine functioning;
  3. = Moderate severity, producing some impairment to routine functioning;
  4. = Severe, causing significant impairment or disability to routine functioning.
Clinical Global Impression-global improvement#CGI-GI# | From enrollment to the end of treatment at 8 weeks
  The Clinical Global Impression (CGI) scale is a comprehensive global assessment instrument. Originally developed by the World Health Organization (WHO) for the International Pilot Study of Schizophrenia (IPSS), it is designed to evaluate clinical treatment outcomes.The Global Improvement (GI) component requires clinicians to assess the degree of improvement or worsening in the patient's condition relative to baseline status. This evaluation compares the patient's current clinical state with their baseline condition at study entry, utilizing an 8-point Likert scale ranging from 0 to 7 for scoring.
Serum Inflammatory Factors | From enrollment to the end of treatment at 8 weeks
  Serum inflammatory factors refer to cytokines, chemokines, acute-phase proteins, and other immune mediators present in bloodstream circulation that participate in systemic inflammatory responses. collection of 5 ml fasting venous blood to measure serum levels of C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-1β (IL-1β), and tumor necrosis fac-tor-α (TNF-α) using enzyme-linked immunosorbent assay (ELISA).

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT07085143/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT07085143/ICF_001.pdf